CLINICAL TRIAL: NCT02797197
Title: Feasibility of Systematic Handgrip Strength (HGS) Testing and Short-term Changes in Muscle Strength in Digestive Cancer Patients Treated by Chemotherapy
Acronym: FIGHTDIGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PO16048
Record Dates: First submitted 2016-06-02; First posted 2016-06-13 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2017-09

CONDITIONS: Handgrip Strength Test; Sarcopenia; Digestive Cancer; Muscle Strength; Chemotherapy
MeSH Terms: conditions — Sarcopenia; Gastrointestinal Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patient undergoing to chemotherapy during 6 months (Experimental)
  Interventions: Procedure: handgrip strength test; Drug: chemotherapy

INTERVENTIONS:
Procedure: handgrip strength test
Drug: chemotherapy

SUMMARY:
Sarcopenia is defined as a loss in skeletal muscle mass and function (strength and/or performance). There is a high prevalence in elderly and in patients with cancer. Several mechanisms are known to explain sarcopenia (inflammation, neurodegenerative process, hormonal disorders, lack of exercise, malnutrition). The consequences were analysed in several studies where sarcopenia appeared to be an independent factor of mortality, and associated with cancer-related fatigue, nosocomial infections, cardio-vascular diseases, and chemotherapy toxicities.

Diagnosis is based on the measure of the muscle mass performing an abdominal computed-tomography (CT) scan, and on the measure of the muscle strength using the handgrip test with a "Jamar®" hydraulic hand dynamometer. CT scan is more invasive and less easy to reach than handgrip test. This test is used to be performing in elderly but not in cancer patients having chemotherapy. Present prospective study explored the feasibility of systematic handgrip strength testing and short-term changes in muscle strength in digestive cancer patients treated by chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with digestive cancer having a chemotherapy and/or biotherapy in the department of Reims
* > 18 years old
* after patient agreement
* linked to social security system

Exclusion Criteria:

* legal guardianship
* < 18 years old
* neuro-muscular issue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
number of patients having at least one handgrip strength test among all hospitalized cancer patients undergoing chemotherapy | 6 months
Evaluation of handgrip test by patients | after 3 months
Evaluation of handgrip test by staff (nurses, interns, students) | 6 months
number of handgrip strength test measures per patient, number of handgrip test measures compared to the number of day hospitalisations, number of patients who had all of the measures, between 50 and 100% of measures, less than 50% of measures | 6 months

SECONDARY OUTCOMES:
to study the association between hand grip strength test and tolerance to chemotherapy | 6 months
to follow the short term evolution of hand grip strength test during 6 months in patients undergoing chemotherapy | 6 months
to study the association between the evolution of hand grip strength test and the evolution of nutritional indices (anthropometric and biologic) | 6 months

REFERENCES:
- [Derived] Perrier M, Ordan MA, Barbe C, Mazza C, Botsen D, Moreau J, Renard Y, Brasseur M, Tailliere B, Regnault P, Bertin E, Bouche O. Dynapenia in digestive cancer outpatients: association with markers of functional and nutritional status (the FIGHTDIGO study). Support Care Cancer. 2022 Jan;30(1):207-215. doi: 10.1007/s00520-021-06416-1. Epub 2021 Jul 12. PMID 34251540
- [Derived] Botsen D, Ordan MA, Barbe C, Mazza C, Perrier M, Moreau J, Brasseur M, Renard Y, Tailliere B, Slimano F, Bertin E, Bouche O. Dynapenia could predict chemotherapy-induced dose-limiting neurotoxicity in digestive cancer patients. BMC Cancer. 2018 Oct 4;18(1):955. doi: 10.1186/s12885-018-4860-1. PMID 30286724